CLINICAL TRIAL: NCT03167918
Title: Liaoning University of Traditional Chinese Medicine
Brief Title: Lung Function in Patients With Early Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Liaoning University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaolin Jiang, Doctor, Liaoning University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140721
Record Dates: First submitted 2017-05-15; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus; Pulmonary Function
Keywords: calcium dobesilate; Xuefuzhuyu Decoction; pulmonary function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Calcium Dobesilate; Metformin; mecobalamin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium dobesilate (Experimental): gave each patient metformin (1000 mg, bid, PO), Mecobalamin Tablets, (0.5 mg bid, PO) and Calcium dobesilate 0.5 g bid, PO
  Interventions: Drug: Calcium Dobesilate; Drug: metformin; Drug: Mecobalamin Tablets
- Xuefuzhuyu Decoction (Experimental): gave each patient metformin (1000 mg, bid, PO), Mecobalamin Tablets, (0.5 mg bid, PO) and Xuefuzhuyu Decoction 100 ml bid，po
  Interventions: Drug: Xuefuzhuyu Decoction; Drug: metformin; Drug: Mecobalamin Tablets
- Xuefuzhuyu Decoction &Calcium dobesilate (Experimental): gave each patient metformin (1000 mg, bid, PO), Mecobalamin Tablets, (0.5 mg bid, PO) and Calcium dobesilate (0.5 g bid, PO)& Xuefuzhuyu Decoction（100 ml bid，po)
  Interventions: Drug: Xuefuzhuyu Decoction & Calcium dobesilate; Drug: metformin; Drug: Mecobalamin Tablets

INTERVENTIONS:
Drug: Calcium Dobesilate — gave each patient 0.5 g bid，
  Arms: Calcium dobesilate
Drug: Xuefuzhuyu Decoction — gave each patient100 ml bid，po
  Arms: Xuefuzhuyu Decoction
Drug: Xuefuzhuyu Decoction & Calcium dobesilate — gave each patient Calcium dobesilate 0.5 g bid，po and Xuefuzhuyu Decoction 100 ml bid，po
  Arms: Xuefuzhuyu Decoction &Calcium dobesilate
Drug: metformin — gave each patient 1000 mg, bid, PO
Drug: Mecobalamin Tablets — gave each patient 0.5 mg bid, PO

SUMMARY:
To investigate the protective effect of calcium dobesilate, Xuefuzhuyu Decoction, calcium dobesilate combined with Xuefuzhuyu Decoction on the early lung function of type 2 diabetes mellitus

DETAILED DESCRIPTION:
Test group and treatment: the patients with type 2 diabetes mellitus were randomly divided into calcium dobesilate group, Xuefuzhuyu Decoction group and combination group. All participants were given hypoglycemic, metformin (1000 mg, bid, PO), Mecobalamin Tablets, nerve nutrition (0.5 mg bid, PO): treatment. Calcium dobesilate group were given hypoglycemic, metformin (500 mg tid, PO), to improve the circular Calcium Dobesilate Capsules (0.5 g bid, PO), Mecobalamin Tablets, nerve nutrition (0.5 mg bid, PO): treatment. Xuefuzhuyu Decoction group was given hypoglycemic, metformin (500 mg tid, PO), to improve the circular Xuefuzhuyu Decoction (100 ml bid, PO), Mecobalamin Tablets, nerve nutrition (0.5 mg bid, PO): treatment. The combined treatment group was given metformin hypoglycemic (500 mg tid, PO), Calcium Dobesilate Capsules, improve circulation (0.5 g bid, PO) + Xuefuzhuyu Decoction (100 ml, bid, PO), Mecobalamin Tablets, nerve nutrition (0.5 mg bid, PO). Before treatment, three groups of patients with blood glucose, oxidation related indicators, retrobulbar hemodynamics and pulmonary function were recorded.

Detection: continuous treatment were observed before and after treatment of the three groups of patients after 24 weeks of fasting blood glucose (FBG), 2 hour postprandial blood glucose (2hPBG), body mass index (BMI), peripheral blood glycated hemoglobin (HbA1c) and related indexes of oxidation, superoxide dismutase (SOD), glutathione peroxidase, Gu Guang (GSH-Px), reactive oxygen species (ROS) activity, malondialdehyde (MDA) concentration and pulmonary function, vital capacity (VC%), forced vital capacity (FVC%), one second forced expiratory flow (FEV1%), peak expiratory flow (PEF%), maximal voluntary ventilation (MVV%), total lung capacity (TCL%) and a second rate (FEV1/FVC%), diffusion capacity of the lung for carbon monoxide (DLCO%), lung volume diffusion capacity of carbon monoxide (DLCO/VA%) changes of the central retinal artery (CRA) and posterior ciliary artery (PCA), eye movement The changes of blood flow velocity and resistance index (RI) of the pulse (AO) systolic and diastolic blood flow were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were diagnosed with type 2 diabetes mellitus according to the guidelines of the American Diabetes Association ;
2. had no history of smoking, pulmonary disease, cold, or pulmonary infection within a two-week period;
3. were not diagnosed with hepatopathy, nephropathy, hyperuricemia, or gastrointestinal disease;
4. were likely to have good compliance and were able to visit our hospital for periodic assessments.

Exclusion Criteria:

1. , type 1 diabetes, pregnant women;
2. there are important organ dysfunction;
3. the need to control blood glucose after insulin injection (poor drug control);
4. the life of patients with irregular or serious addiction (alcoholism),
5. poor compliance and compliance;
6. the experiment of drug intolerance (severe allergic reaction 6);
7. hypertension and hyperuricemia;
8. and nearly two weeks colds, pneumonia and other respiratory diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in pulmonary function parameters | 26 weeks
  The primary endpoints were the between-group differences in the changes in pulmonary function parameters between pretherapy and posttreatment

SECONDARY OUTCOMES:
Changes in glycosylated hemoglobinA1c, fasting plasma glucose, 2-hour postprandial blood glucose, | 26 weeks
  The secondary endpoints were changes from baseline to week 26 in glycosylated hemoglobinA1c, fasting plasma glucose, 2-hour postprandial blood glucose,. The tertiary endpoints were the changes from baseline to week 26 in blood-fat

OTHER OUTCOMES:
Changes in blood-fat in Systolic blood pressure,Diastolic blood pressure, and blood-fat | 26 weeks
  The quartus endpoints were the changes from baseline to week 26 in Systolic blood pressure,Diastolic blood pressure, and blood-fat
Changes in retrobulbar hemodynamics (RI) | 26 weeks
  The fifth endpoints were the changes from baseline to week 26 in retrobulbar hemodynamics (RI) in the bilateral central retinal artery,posterior ciliary artery, endarteria ophthalmica.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-lin Jiang, Principal Investigator — Liaoning University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No